CLINICAL TRIAL: NCT05910892
Title: The Effect of Aromatherapy on the Incidence and Severity of Post Procedure Pain and Discomfort in Patients
Brief Title: Aromatherapy and Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contract was never finalized and UW GCA closed the study due to lack of funding and activity.
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Heather Tick, Clinical Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00007869
Record Dates: First submitted 2023-04-29; First posted 2023-06-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Intramuscular Stimulation Therapy; Trigger Point Injections; Aromatherapy
MeSH Terms: conditions — Chronic Pain | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aromatherapy before treatment (Active Comparator): Subject receives aromatherapy before IMS treatment or trigger point injection
  Interventions: Drug: Aromatherapy packet
- Placebo before treatment (Placebo Comparator): Subject receives placebo before IMS treatment or trigger point injection
  Interventions: Drug: Placebo packet

INTERVENTIONS:
Drug: Aromatherapy packet — 5 deep breaths from packet prior to treatment
  Other Names: Aromatherapy
  Arms: Aromatherapy before treatment
Drug: Placebo packet — 5 deep breaths from packet prior to treatment
  Other Names: Placebo
  Arms: Placebo before treatment

SUMMARY:
Effect of aromatherapy on pain and discomfort in patients who are receiving intramuscular stimulation therapy or trigger point injections for chronic pain.

DETAILED DESCRIPTION:
The study will explore the effect of aromatherapy on pain and discomfort in patients who are receiving intramuscular stimulation therapy or trigger point injections for chronic pain. This will be a blinded study where patients will act as their own control over two treatment visits. On one visit patient will be exposed to either the aromatherapy or a placebo. On their second visit patients will be exposed to the other compound. The study will collect demographic data, pain intensity and affect, and catastrophizing information.

ELIGIBILITY:
Inclusion Criteria:

* Have received at least one (1) prior IMS or trigger point injection treatment with researcher
* 18 years of age or older
* English language speaker
* has completed Pain Tracker (clinic standard of care) questionnaire prior to study visit
* any analgesic medication taken must be consistent for both sessions

Exclusion Criteria:

* Non-English language speaker
* Age <18
* Allergy to essential oils
* Asthmatic
* Patient unable to self-administer aromatherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Acute Pain | Immediately after the Procedure
  Examine the change in Acute Pain associated with two identical procedures involving muscle with either an aromatherapy intervention or control intervention. With each patient being their own control, patients will rate their acute pain immediately after the procedure on a 0-10 scale (0=No pain and 10=Pain as bad as you can imagine).

SECONDARY OUTCOMES:
Change in Overall Experience | Immediately after the Procedure
  Examine the change in Overall Experience of pain with two identical procedures involving muscle with either an aromatherapy intervention or control intervention. With each patient being their own control, patients will rate their overall experience of pain after the procedure on a 0-10 scale (0=No pain and 10=Pain as bad as you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Tick, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No